CLINICAL TRIAL: NCT00000145
Title: Age-Related Eye Disease Study (AREDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: John Paul SanGiovanni, Sc.D., National Eye Institute
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEI-44; NCT00001312 (obsolete NCT alias)
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Macular Degeneration; Cataract; Lens Opacities
Keywords: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Cataract | interventions — Antioxidants; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Antioxidants
  Interventions: Dietary Supplement: Antioxidants
- 2 (Experimental): Zinc
  Interventions: Dietary Supplement: Zinc
- 3 (Experimental): Antioxidants and zinc
  Interventions: Dietary Supplement: Antioxidants and zinc
- 4 (No Intervention)

INTERVENTIONS:
Dietary Supplement: Antioxidants — 500 milligrams vitamin C; 400 IUs vitamin E; 15 milligrams beta-carotene
  Arms: 1
Dietary Supplement: Zinc — 80 milligrams zinc oxide; 2 milligrams of cupric oxide
  Arms: 2
Dietary Supplement: Antioxidants and zinc — 500 milligrams vitamin C; 400 IUs vitamin E; 15 milligrams beta-carotene; 80 milligrams zinc oxide; 2 milligrams of cupric oxide
  Arms: 3

SUMMARY:
To assess the clinical course, prognosis, and risk factors of age-related macular degeneration (AMD) and cataract.

To evaluate, in randomized clinical trials, the effects of pharmacologic doses of (1) antioxidants and zinc on the progression of AMD and (2) antioxidants on the development and progression of lens opacities.

DETAILED DESCRIPTION:
AMD and cataract are the leading causes of visual impairment and blindness in the United States. Based on many clinical studies, it is apparent that the frequency of both diseases increases dramatically after age 60. Although excellent treatments for cataract are available, there are no equivalent treatments for AMD. As the average lifespan of our population increases, the number of people who develop AMD will increase dramatically in the years ahead. Unless successful means of prevention or treatment are developed, blindness from AMD -- and its importance as a public health problem -- will increase.

Neither the etiology nor the natural history of AMD or cataract is known. Epidemiologic studies suggest that a number of risk factors may be associated with AMD and cataract, but the strength of the evidence in support of these hypotheses varies. Possibly associated with AMD are personal characteristics, such as age, race, height, family history, and strength of hand grip; ocular characteristics, such as hyperopia and color of iris; and cardiovascular diseases, smoking, lung infections, and chemical exposures. Clinical and laboratory studies suggest the following factors may be associated with progression of AMD: drusen type, choroidal vascular diseases, and photic injury.

Epidemiologic studies of cataract suggest that associated risk factors may include personal characteristics, such as age, sex, race, occupation, and educational status; ocular characteristics, such as iris color; and diabetes mellitus, hypertension, drug exposure, smoking, and sunlight exposure. Animal studies and observational epidemiologic studies suggest that deficiencies in vitamins C and E, carotenoids, and the trace elements zinc and selenium also may be associated with the development of the two diseases, especially cataract. Although surgical treatment to remove cataract is very effective, cataract surgery carries risks, as does any other surgery. Therefore, many research efforts focus on preventing or slowing cataract development, as well as on determining the causes of cataract formation.

The Age-Related Eye Disease Study (AREDS) is a major research program to improve our understanding of the predisposing factors, clinical course, and prognostic factors of AMD and cataract. Eligible patients are randomized to treatment with placebo, antioxidants, zinc, or antioxidants plus zinc, and are followed for a minimum of 5 years.

ELIGIBILITY:
Men and women between the ages of 55 and 80 years whose macular status ranges from no evidence of AMD in either eye to relatively severe disease with vision loss in one eye but good vision in the fellow eye (20/30 or better) are eligible for the study provided that their ocular media are clear enough to allow good fundus photography.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4757 (Actual)
Dates: Start 1990-09; Primary Completion 2001-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Progression of age-related macular degeneration
Progression of lens opacity (cataract)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y. Chew, MD, Principal Investigator — National Eye Institute (NEI)

REFERENCES:
- [Background] Age-Related Eye Disease Study Research Group. The Age-Related Eye Disease Study system for classifying age-related macular degeneration from stereoscopic color fundus photographs: the Age-Related Eye Disease Study Report Number 6. Am J Ophthalmol. 2001 Nov;132(5):668-81. doi: 10.1016/s0002-9394(01)01218-1. PMID 11704028
- [Background] Age-Related Eye Disease Study Research Group. The age-related eye disease study (AREDS) system for classifying cataracts from photographs: AREDS report no. 4. Am J Ophthalmol. 2001 Feb;131(2):167-75. doi: 10.1016/s0002-9394(00)00732-7. PMID 11228291
- [Background] Age-Related Eye Disease Study Research Group. The Age-Related Eye Disease Study (AREDS): design implications. AREDS report no. 1. Control Clin Trials. 1999 Dec;20(6):573-600. doi: 10.1016/s0197-2456(99)00031-8. PMID 10588299
- [Background] Clemons TE, Chew EY, Bressler SB, McBee W; Age-Related Eye Disease Study Research Group. National Eye Institute Visual Function Questionnaire in the Age-Related Eye Disease Study (AREDS): AREDS Report No. 10. Arch Ophthalmol. 2003 Feb;121(2):211-7. doi: 10.1001/archopht.121.2.211. PMID 12583787
- [Background] Bressler NM, Bressler SB, Congdon NG, Ferris FL 3rd, Friedman DS, Klein R, Lindblad AS, Milton RC, Seddon JM; Age-Related Eye Disease Study Research Group. Potential public health impact of Age-Related Eye Disease Study results: AREDS report no. 11. Arch Ophthalmol. 2003 Nov;121(11):1621-4. doi: 10.1001/archopht.121.11.1621. PMID 14609922
- [Background] Lindblad AS, Clemons TE. Responsiveness of the National Eye Institute Visual Function Questionnaire to progression to advanced age-related macular degeneration, vision loss, and lens opacity: AREDS Report no. 14. Arch Ophthalmol. 2005 Sep;123(9):1207-14. doi: 10.1001/archopht.123.9.1207. PMID 16157800
- [Background] Rankin MW, Clemons TE, McBee WL. Correlation analysis of the in-clinic and telephone batteries from the AREDS cognitive function ancillary study. AREDS Report No. 15. Ophthalmic Epidemiol. 2005 Aug;12(4):271-7. doi: 10.1080/09286580591003815. PMID 16033748
- [Background] Davis MD, Gangnon RE, Lee LY, Hubbard LD, Klein BE, Klein R, Ferris FL, Bressler SB, Milton RC; Age-Related Eye Disease Study Group. The Age-Related Eye Disease Study severity scale for age-related macular degeneration: AREDS Report No. 17. Arch Ophthalmol. 2005 Nov;123(11):1484-98. doi: 10.1001/archopht.123.11.1484. PMID 16286610
- [Background] Ferris FL, Davis MD, Clemons TE, Lee LY, Chew EY, Lindblad AS, Milton RC, Bressler SB, Klein R; Age-Related Eye Disease Study (AREDS) Research Group. A simplified severity scale for age-related macular degeneration: AREDS Report No. 18. Arch Ophthalmol. 2005 Nov;123(11):1570-4. doi: 10.1001/archopht.123.11.1570. PMID 16286620
- [Background] Sperduto RD, Ferris FL 3rd, Kurinij N. Do we have a nutritional treatment for age-related cataract or macular degeneration? Arch Ophthalmol. 1990 Oct;108(10):1403-5. doi: 10.1001/archopht.1990.01070120051026. No abstract available. PMID 2222272
- [Result] Age-Related Eye Disease Study Research Group. The effect of five-year zinc supplementation on serum zinc, serum cholesterol and hematocrit in persons randomly assigned to treatment group in the age-related eye disease study: AREDS Report No. 7. J Nutr. 2002 Apr;132(4):697-702. doi: 10.1093/jn/132.4.697. PMID 11925463
- [Result] Age-Related Eye Disease Study Research Group. Risk factors associated with age-related nuclear and cortical cataract : a case-control study in the Age-Related Eye Disease Study, AREDS Report No. 5. Ophthalmology. 2001 Aug;108(8):1400-8. doi: 10.1016/s0161-6420(01)00626-1. PMID 11470690
- [Result] Age-Related Eye Disease Study Research Group. Risk factors associated with age-related macular degeneration. A case-control study in the age-related eye disease study: Age-Related Eye Disease Study Report Number 3. Ophthalmology. 2000 Dec;107(12):2224-32. doi: 10.1016/s0161-6420(00)00409-7. PMID 11097601
- [Result] Age-Related Eye Disease Study Research Group. The Age-Related Eye Disease Study: a clinical trial of zinc and antioxidants--Age-Related Eye Disease Study Report No. 2. J Nutr. 2000 May;130(5S Suppl):1516S-9S. doi: 10.1093/jn/130.5.1516S. PMID 10801969
- [Result] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E and beta carotene for age-related cataract and vision loss: AREDS report no. 9. Arch Ophthalmol. 2001 Oct;119(10):1439-52. doi: 10.1001/archopht.119.10.1439. PMID 11594943
- [Result] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol. 2001 Oct;119(10):1417-36. doi: 10.1001/archopht.119.10.1417. PMID 11594942
- [Result] Yaffe K, Clemons TE, McBee WL, Lindblad AS; Age-Related Eye Disease Study Research Group. Impact of antioxidants, zinc, and copper on cognition in the elderly: a randomized, controlled trial. Neurology. 2004 Nov 9;63(9):1705-7. doi: 10.1212/01.wnl.0000142969.19465.8f. PMID 15534261
- [Result] Clemons TE, Kurinij N, Sperduto RD; AREDS Research Group. Associations of mortality with ocular disorders and an intervention of high-dose antioxidants and zinc in the Age-Related Eye Disease Study: AREDS Report No. 13. Arch Ophthalmol. 2004 May;122(5):716-26. doi: 10.1001/archopht.122.5.716. PMID 15136320
- [Result] Clemons TE, Rankin MW, McBee WL; Age-Related Eye Disease Study Research Group. Cognitive impairment in the Age-Related Eye Disease Study: AREDS report no. 16. Arch Ophthalmol. 2006 Apr;124(4):537-43. doi: 10.1001/archopht.124.4.537. PMID 16606880
- [Result] Clemons TE, Milton RC, Klein R, Seddon JM, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Risk factors for the incidence of Advanced Age-Related Macular Degeneration in the Age-Related Eye Disease Study (AREDS) AREDS report no. 19. Ophthalmology. 2005 Apr;112(4):533-9. doi: 10.1016/j.ophtha.2004.10.047. PMID 15808240
- [Result] SanGiovanni JP, Chew EY, Clemons TE, Davis MD, Ferris FL 3rd, Gensler GR, Kurinij N, Lindblad AS, Milton RC, Seddon JM, Sperduto RD; Age-Related Eye Disease Study Research Group. The relationship of dietary lipid intake and age-related macular degeneration in a case-control study: AREDS Report No. 20. Arch Ophthalmol. 2007 May;125(5):671-9. doi: 10.1001/archopht.125.5.671. PMID 17502507
- [Result] Milton RC, Sperduto RD, Clemons TE, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Centrum use and progression of age-related cataract in the Age-Related Eye Disease Study: a propensity score approach. AREDS report No. 21. Ophthalmology. 2006 Aug;113(8):1264-70. doi: 10.1016/j.ophtha.2006.02.054. PMID 16877067
- [Result] Age-Related Eye Disease Study Research Group; SanGiovanni JP, Chew EY, Clemons TE, Ferris FL 3rd, Gensler G, Lindblad AS, Milton RC, Seddon JM, Sperduto RD. The relationship of dietary carotenoid and vitamin A, E, and C intake with age-related macular degeneration in a case-control study: AREDS Report No. 22. Arch Ophthalmol. 2007 Sep;125(9):1225-32. doi: 10.1001/archopht.125.9.1225. PMID 17846363
- [Result] SanGiovanni JP, Chew EY, Agron E, Clemons TE, Ferris FL 3rd, Gensler G, Lindblad AS, Milton RC, Seddon JM, Klein R, Sperduto RD; Age-Related Eye Disease Study Research Group. The relationship of dietary omega-3 long-chain polyunsaturated fatty acid intake with incident age-related macular degeneration: AREDS report no. 23. Arch Ophthalmol. 2008 Sep;126(9):1274-9. doi: 10.1001/archopht.126.9.1274. PMID 18779490
- [Result] Sperduto RD, Clemons TE, Lindblad AS, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Cataract classification using serial examinations in the age-related eye disease study: age-related eye disease study report no. 24. Am J Ophthalmol. 2008 Mar;145(3):504-8. doi: 10.1016/j.ajo.2007.10.024. Epub 2008 Jan 16. PMID 18201681
- [Derived] Toulouie S, Chang S, Pan J, Snyder K, Yiu G. Relationship of Retinal Vessel Caliber with Age-Related Macular Degeneration. J Ophthalmol. 2022 Jul 31;2022:8210599. doi: 10.1155/2022/8210599. eCollection 2022. PMID 35957743
- [Derived] Snyder K, Yazdanyar A, Mahajan A, Yiu G. Association Between the Cilioretinal Artery and Choroidal Neovascularization in Age-Related Macular Degeneration: A Secondary Analysis From the Age-Related Eye Disease Study. JAMA Ophthalmol. 2018 Sep 1;136(9):1008-1014. doi: 10.1001/jamaophthalmol.2018.2650. PMID 29978186
- [Derived] Chiu CJ, Klein R, Milton RC, Gensler G, Taylor A. Does eating particular diets alter the risk of age-related macular degeneration in users of the Age-Related Eye Disease Study supplements? Br J Ophthalmol. 2009 Sep;93(9):1241-6. doi: 10.1136/bjo.2008.143412. Epub 2009 Jun 9. PMID 19508997